CLINICAL TRIAL: NCT06810414
Title: Feasibility, Acceptability, and Preliminary Efficacy of an Expectancy Challenge Intervention for Food and Alcohol Disturbance Among College Students
Brief Title: Evaluation of an Expectancy Challenge Intervention for Food and Alcohol Disturbance Among College Students
Acronym: FAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wyoming (Other)
Responsible Party: Principal Investigator, Katherine Berry, Clinical Psychology Doctoral Candidate, University of Wyoming
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2024-467
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: College Drinking; Disordered Eating
Keywords: food and alcohol disturbance; drunkorexia; college drinking; disordered eating; expectancy challenge
MeSH Terms: conditions — Alcohol Drinking in College | interventions — Food; Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAD Expectancy Challenge Condition (Experimental): Participants in the experimental condition will be delivered the FAD expectancy challenge intervention.
  Interventions: Behavioral: Food and alcohol disturbance expectancy challenge
- Disordered Eating Psychoeducation (No Intervention): Participants in the control condition will receive psychoeducation on disordered eating behaviors, with only a brief mention of FAD, and excluding any discussion of expectancies and consequences.

INTERVENTIONS:
Behavioral: Food and alcohol disturbance expectancy challenge — The intervention will focus on strengthening negative FAD expectancies and weakening positive FAD expectancies.
  Arms: FAD Expectancy Challenge Condition

SUMMARY:
This study aims to create and test an intervention that helps college students re-evaluate their beliefs about food and alcohol disturbance (FAD) and, in turn, reduce how often they engage in it or intend to in the future. The main questions it aims to answer are:

1. Does the intervention help students have less positive beliefs about the effects of FAD and more negative beliefs about its effects?
2. If college students' beliefs about FAD change, does that lead them to engage in it less often or plan to do it less?
3. Will college students who engage in FAD sign up for the study, complete it, and feel that the intervention is helpful and valuable?

Participants will take part in one 2-hour in-person laboratory-based study session where they will fill out surveys, learn about FAD, and engage in exercises designed to challenge their existing beliefs about it. They will also complete a follow-up survey online one month after their in-person study visit.

DETAILED DESCRIPTION:
Food and alcohol disturbance (FAD) is the use of any compensatory behavior (e.g., caloric restriction) within the context of a drinking episode for the purpose of 1) compensating for alcohol-related calories and/or 2) enhancing the effects of alcohol. FAD occurs at alarmingly high rates among undergraduates and is associated with a myriad of deleterious consequences. Expectancy effects (i.e., beliefs regarding the anticipated outcomes of a behavior) have been shown to influence the initiation and maintenance of alcohol and disordered eating behaviors. Prior work suggests that expectancies for these behaviors can be modified via expectancy challenges (i.e., ECs; interventions that aim to undermine expectancies by providing learning opportunities that demonstrate the discrepancy between the actual versus perceived effects of a behavior). An EC has never been applied to FAD. However, given that FAD is comprised of both alcohol and disordered eating behaviors, and preliminary work suggests that FAD expectancies share some similarities with alcohol and restriction expectancies, it is likely that an EC could be similarly applied to FAD. Thus, the purpose of the proposed project is to develop an effective and acceptable EC designed to modify FAD expectancies and reduce FAD among undergraduates, informed by the alcohol EC literature.

Participants will be randomized to a 120-minute in-person non-experiential (i.e., no alcohol administration) EC designed to undermine FAD expectancies (experimental group) or a control group. To make existing expectancies salient, the EC will include audio recordings of reported FAD expectancies from students who engaged in FAD in my preliminary qualitative work (Berry & Looby, 2024). Participants will then engage in discussions to evaluate whether these effects are pharmacological or perceived. The intervention will also provide psychoeducation on expectancies, FAD, alcohol, and the effects of compensatory behaviors on weight, which will prompt participants to reevaluate their extant expectancies. This will be followed by a reflective writing exercise to allow participants to further elaborate on any changes to their challenged expectancies. FAD expectancies will be assessed at baseline, immediately post-intervention, and one-month follow-up. FAD frequency will be assessed at baseline and follow-up. Additionally, participants in the experimental group will provide feedback on the intervention's acceptability and feasibility post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Must be between the ages of 18 and 25
2. Must report engaging in FAD at least two times over the past month

Exclusion Criteria:

1. They have a current or past history of receiving psychological treatment for their alcohol use and/or eating behaviors
2. They are currently trying to reduce their drinking

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-02-24 (Estimated); Primary Completion 2026-05-08 (Estimated); Study Completion 2026-05-08 (Estimated)

PRIMARY OUTCOMES:
Food and Alcohol Disturbance Expectancy Questionnaire | This measure will be administered to all participants at baseline, immediately post-intervention, and at the study's one-month follow-up
  The Food and Alcohol Disturbance Expectancy Questionnaire is a 30-item self-report questionnaire that assesses positive and negative expectancies for FAD. Participants will be asked to indicate the extent to which they believe or expect each FAD-related outcome to occur if they engaged in FAD, using a five-point scale from 0 (Strongly Disagree) to 5 (Strongly Agree). Scores on each factor will be summed and averaged, with higher scores indicating stronger expectancies.
Food and Alcohol Disturbance Intentions Questions | This measure will be administered to all participants at baseline, immediately post-intervention, and at the study's one-month follow-up
  Two questions will be used to assess intentions to engage in FAD for both caloric compensation and alcohol enhancement motives. Items will be rated on a scale from 0 (Very unlikely) to 10 (Very likely), with higher scores indicating greater intentions to engage in FAD.
College Eating and Drinking Behaviors Scale | This measure will be administered at baseline and at the one-month follow-up
  The CEDBS is a 21-item questionnaire that measures the frequency of past-month FAD. Items are rated on a scale from 1 (Never) to 6 (Always), with higher scores indicating more frequent FAD.
Food and Alcohol Disturbance Timeline Followback | This measure will be administered at baseline and at the one-month follow-up
  This measure will assess past-month FAD frequency, including FAD motives and compensatory behaviors. The number of days that participants reported engaging in FAD will be summed, with higher scores indicating more frequent FAD.

SECONDARY OUTCOMES:
Brief Young Adult Alcohol Consequences Questionnaire | This measure will be administered at baseline and at the one-month follow-up
  The Brief Young Adult Alcohol Consequences Questionnaire is a 24-item self-reported questionnaire that assesses past-month alcohol-related negative consequences using a dichotomous "Yes" or "No" response item format. A composite score indicating how many consequences participants experienced will be created by summing the number of alcohol problems reported. Higher scores will represent greater alcohol consequences.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Berry, MS, Principal Investigator — University of Wyoming; Alison Looby, PhD, Study Chair — University of Wyoming
Locations (1):
- University of Wyoming, Laramie, Wyoming, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berry KA, Looby A. "If You Don't Eat, You Can Get Drunk Faster": A Qualitative Investigation of Food and Alcohol Disturbance (FAD) Expectancies. Subst Use Misuse. 2024;59(11):1647-1655. doi: 10.1080/10826084.2024.2369161. Epub 2024 Jun 25. PMID 38918931
- [Background] Berry KA, Choquette EM, Looby A, Rancourt D. Unification of the food and alcohol disturbance literature: A systematic review. Clin Psychol Rev. 2024 Nov;113:102486. doi: 10.1016/j.cpr.2024.102486. Epub 2024 Aug 14. PMID 39168054
- [Background] Shepherd CB, Berry KA, Ye X, Li K. Food and alcohol disturbance among US college students: a mixed methods scoping review. J Am Coll Health. 2023 Aug-Sep;71(6):1715-1731. doi: 10.1080/07448481.2021.1947300. Epub 2021 Jul 22. PMID 34292851

DOCUMENTS (1):
  • Informed Consent Form (2024-12-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT06810414/ICF_001.pdf